CLINICAL TRIAL: NCT05154266
Title: Effectiveness of 'Taking it Further' (TiF) Programme Compared to Waitlist Control in the Promotion of Well-being and Mental Health: A Randomised Controlled Trial With Graduates of MBCT and MBSR
Brief Title: Effectiveness of 'Taking it Further' (TiF) Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mind and Life Europe (Unknown)
Responsible Party: Principal Investigator, ProfessorWillemKuyken, Professor, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TiF2021; 2020EVA-Maloney, Shannon (Other Grant/Funding Number: Mind and Life Europe)
Record Dates: First submitted 2021-11-29; First posted 2021-12-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Mindfulness
Keywords: Mindfulness-Based Cognitive Therapy; Mechanism; Mediator; Well-being; Mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Wait-list control
Who Masked: Outcomes Assessor
Masking Description: The experimenter was unaware of who was allocated to the treatment or control group during data collection and analysis. A researcher external to data collection and analysis was in charge of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Programme (Experimental): Participants randomized to the mindfulness programme were invited to complete a twelve-week programme called 'Taking it Further'.
  Interventions: Behavioral: Taking it Further
- Waitlist Control (No Intervention): Participants randomized to the waitlist control were asked to carry on as usual and were offered the Taking it Further course at a later time. No data was collected when the waitlist control group took part in the TiF programme.

INTERVENTIONS:
Behavioral: Taking it Further — This programme is offered to individuals who have already completed a Mindfulness-Based Cognitive Therapy (MBCT) or Mindfulness-Based Stress Reduction Programme (MBSR). In this programme, participants explore weekly themes (i.e. 'Responding not reacting' and 'Taking care of ourselves, taking care of others'). These themes reinforce the learning from the eight-week MBCT/MBSR courses whilst also providing new learning opportunities. The programme makes some of the dimensions that are implicit in MBCT/MBSR more explicit; for example, the cultivation of attitudes of mindfulness (such as equanimity, joy, and kindness). These attitudes of mindfulness require a foundational mindfulness practice and thus this is an additive learning theme from traditional MBCT/MBSR programmes.
  Arms: Mindfulness Programme

SUMMARY:
Meta-analyses have demonstrated that mindfulness-based programmes are more effective than no treatment across different populations and desired outcomes yet there is limited evidence on how to sustain these benefits beyond the traditional eight-week courses. The 'Taking it Further' (TiF) programme was developed by the University of Oxford Mindfulness Centre to help reinforce and deepen one's mindfulness practice to promote well-being and mental health for life. The proposed study aims to evaluate the effectiveness of this programme in graduates of MBCT/MBSR on well-being and mental health outcomes and explore the mediators (i.e. mindfulness, decentring, and self-compassion) through which this programme has an effect over the course of twelve weeks using a randomised controlled trial with a waitlist control. The planned research is part of an overall effort to optimize treatment effects and the long-term effectiveness of mindfulness-based programmes.

DETAILED DESCRIPTION:
Participants that expressed an interest in taking part in the study were screened for research inclusion/exclusion criteria and for course suitability. Research inclusion/exclusion was assessed by the lead researcher whereas course suitability was assessed jointly by the lead researcher and a trained mindfulness teacher at the Oxford Mindfulness Centre (OMC). Eligible participants were invited to complete baseline measures that assessed the primary outcome and mediator (well-being and mindfulness respectively) around two weeks before the start date and then again around one week before the start date to establish a stable baseline. For one of these online questionnaires, participants were instructed to complete an online orientation video to ensure continued eligibility. Within a few days of the start date, participants were randomised to the treatment (online TiF programme) or wait-list control group. One day before the start date, all participants were invited to complete a battery of questionnaires which assessed the outcome measures (well-being, psychological quality of life, depression, anxiety), mediator measures (mindfulness, self-compassion, decentring), and an additional measure regarding perceived expectations about the mindfulness course. Participants were then invited to complete a battery of questionnaires at weeks 4, 8, and 12 (post-intervention). For the battery of questionnaires for weeks 4 and 8, participants completed the same measures assessed at baseline with additional questions that assessed: the amount of practice, quality of practice, side effects of practice, and overall experience. For week 12 (post-intervention), participants completed the same measures as weeks 4 and 8 with additional questions that assessed the perceived credibility of the mindfulness programme, perceived quality of mindfulness teaching, and potential harm. Data collection was divided into two phases, with the first phase running from June-September and the second phase running from October-December 2021. The TiF courses were run online and the surveys themselves were also administered online.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Has access to computer for online mindfulness sessions and assessments
* Participants who have completed an MBSR and/or MBCT course in the past

Exclusion Criteria:

* Has taken TiF programme prior to the start of the study
* Has completed a mindfulness programme that does not fit within the parameters of a formal mindfulness-based programme.
* Those that have recently experienced a traumatic event or bereavement and/or has been abusing substances to manage stress and/or has been harming themselves recently
* Participants on mindfulness teacher training pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Change in Well-being | Pre-intervention (~2 weeks and 1 week before Week 0), Week 0, Week 4, Week 8, Week 12 (Post-intervention)
  To explore the effects of the TiF programme on well-being over time, the 14-item Warwick-Edinburgh Mental Well-being Scale (WEMWBS) will be used.

SECONDARY OUTCOMES:
Change in Mindfulness | Pre-intervention (~2 weeks and 1 week before Week 0), Week 0, Week 4, Week 8, Week 12 (Post-intervention)
  To explore the effects of the TiF programme on mindfulness over time, the Five Facet Mindfulness Questionnaire Short-Form (FFMQ-15) will be used.
Change in Psychological Quality of Life | Week 0, Week 4, Week 8, Week 12 (Post-intervention)
  To investigate the effects of the TiF programme on psychological quality of life over time, the 6-item psychological domain of the WHO-QOL-BREF questionnaire will be used.
Change in Depression | Week 0, Week 4, Week 8, Week 12 (Post-intervention)
  To evaluate the effects of the TiF programme on symptoms of depression over time, the 9-item Patient Health Questionnaire (PHQ-9) will be used.
Change in Anxiety | Week 0, Week 4, Week 8, Week 12 (Post-intervention)
  To investigate the effects of the TiF programme on anxiety over time, the 7-item Generalized Anxiety Disorder (GAD-7) will be used.
Change in Self-compassion | Week 0, Week 4, Week 8, Week 12 (Post-intervention)
  To explore the effects of the TiF programme on self-compassion over time, the 12-item Self-Compassion Scale Short-Form (SCS-SF) will be used.
Change in Decentring | Week 0, Week 4, Week 8, Week 12 (Post-intervention)
  To explore the effects of the TiF programme on decentring over time, the 11-item Experiences Questionnaire (EQ) will be used.

OTHER OUTCOMES:
Amount of mindfulness practice | Week 4, Week 8, Week 12 (Post-intervention)
  The amount of mindfulness practice will be meausured using daily journal logs and participants will be asked about the amount of practice every four weeks retrospectively.
Change in quality of mindfulness practice | Week 4, Week 8, Week 12 (Post-intervention)
  To assess the quality of mindfulness practice, the Practice Quality-Mindfulness (PQ-M) questionnaire will be used.
Change in side effects of mindfulness practice | Week 4, Week 8, Week 12 (Post-intervention)
  Participants will be asked about their experience (including potential side effects of mindfulness practice) across a twelve-week period using open-ended questions.
Perceived expectations | Week 0
  Participants will be asked about perceived expectations about the TiF programme before they took part.
Perceived credibility | Week 12 (Post-intervention)
  Participants will be asked about perceived credibility of the TiF programme after they completed the programme.
Perceived quality of teaching | Week 12 (Post-intervention)
  Participants allocated to treatment will be asked about perceived quality of teaching received during the TiF programme.
Potential harm | Week 12 (Post-intervention)
  Participants will be asked about perceived harm over the course of twelve weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Willem Kuyken, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montero-Marin J, Farley ER, Maloney S, Crane R, D'Alton P, Eldridge R, Giommi F, Griffith G, Hecht FM, Hinze V, Loucks EB, Strauss C, Taylor L, Baer R, Kuyken W. Participants' Perspective on the Competence of Mindfulness-Based Interventions Teaching: Development and Validation of the Mindfulness-Based Interventions-Participants' Assessment of Teaching (MBI:PAT) Questionnaire. Mindfulness (N Y). 2025;16(10):2825-2844. doi: 10.1007/s12671-025-02668-8. Epub 2025 Sep 3. PMID 41322157
- [Derived] Maloney S, Montero-Marin J, Kuyken W. Mindfulness-Based Cognitive Therapy-Taking it Further (MBCT-TiF) compared to Ongoing Mindfulness Practice (OMP) in the promotion of well-being and mental health: A randomised controlled trial with graduates of MBCT and MBSR. Behav Res Ther. 2024 Feb;173:104478. doi: 10.1016/j.brat.2024.104478. Epub 2024 Jan 6. PMID 38244384
- [Derived] Maloney S, Montero-Marin J, Kuyken W. Pathways to mental well-being for graduates of mindfulness-based cognitive therapy (MBCT) and mindfulness-based stress reduction (MBSR): A mediation analysis of an RCT. Psychother Res. 2024 Nov;34(8):1162-1173. doi: 10.1080/10503307.2023.2269299. Epub 2023 Nov 6. PMID 37931304